CLINICAL TRIAL: NCT05901597
Title: Refractive Accuracy of Argos in Conjunction With the Alcon Vision Suite Following Implantation of Presbyopia Correcting IOLs
Status: Recruiting | Type: Observational
Sponsor: Valley Laser Eye Centre (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JB-23-01
Record Dates: First submitted 2023-06-02; First posted 2023-06-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Clareon PanOptix and AcrySof Vivity IOL implantation Alcon Vision Suite and Argos biometer — Clareon PanOptix and AcrySof Vivity IOL implantation Alcon Vision Suite and Argos biometer

SUMMARY:
The objective is to assess refractive accuracy of the Alcon Vision Suite (with Argos biometer) following Clareon PanOptix and AcrySof Vivity IOL implantation.

DETAILED DESCRIPTION:
This study is a single-arm, observational study of refractive accuracy of the Alcon Vision Suite (with Argos biometer) following Clareon PanOptix and AcrySof Vivity IOL implantation. Subjects will be assessed at preoperatively, operatively, and 10 weeks post-operatively. Clinical evaluations will include measurement of monocular and binocular visual acuity, manifest refraction, and questionnaires will also be administered.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Age-related cataract surgery (or RLE) patients that select Clareon PanOptix or AcrySof Vivity IOL.
* Gender: Males and Females.
* Age: 45 or older.
* Patients motivated to increase spectacle independence with relatively low incidence of visual phenomena.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error).

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Ocular comorbidity (any previous ocular surgery, any signs of retinal disease, or glaucoma etc.) that might hamper post-operative visual acuity.
* Irregular corneal astigmatism and keratoconus.
* Post refractive eyes (i.e. LASIK or PRK or SMILE).
* Patients with physical or intellectual disability (e.g. Down's Syndrome, Parkinson's Disease; unable to fixate).
* Angle Kappa/chord mu ≥0.6.
* Higher order corneal aberrations: > 0.6 total RMS, >0.3 coma, >0.3 trefoil (to exclude irregular corneas).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with age-related cataracts (or refractive lens exchange), and a motivation for spectacle independence.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Monocular refractive target accuracy | 10 Weeks postoperative
  Percentage of subjects within predicted postoperative spherical equivalent of ± 0.5 D.

SECONDARY OUTCOMES:
Prediction error | 10 Weeks postoperative
  Percentage of eyes within prediction errors (PE) of ± 0.25D, 0.75D, 1.0D
Mean absolute prediction error | 10 Weeks postoperative
Median absolute prediction error | 10 Weeks postoperative
Uncorrected monocular visual acuity | 10 Weeks postoperative
  at distance (6m), intermediate (60cm), and near (40cm)
Distance corrected monocular visual acuity | 10 Weeks postoperative
  at distance (6m), intermediate (60cm), and near (40cm)
Manifest refraction | 10 Weeks postoperative
Back-calculated Residual Astigmatism (BRA) | 10 Weeks postoperative
  using preoperative cylinder power (for toric IOLs)

OTHER OUTCOMES:
Uncorrected binocular visual acuity | 10 Weeks postoperative
  at distance (6m), intermediate (60cm), and near (40cm)
Satisfaction questionnaire | 10 Weeks postoperative
  The Intraocular Lens Satisfaction questionnaire (IOLSAT). Lower scores indicate higher spectacle independence and satisfaction.
Visual disturbances questionnaire | 10 Weeks postoperative
  Questionnaire for Visual Disturbances (QUVID). Lower scores indicate less frequent, severe, or bothersome visual disturbances.
Percentage of cases in which IA IOL power recommendation differed from preop calculation | 10 Weeks postoperative

CONTACTS AND LOCATIONS:
Overall Officials: John Blaylock, MD, Principal Investigator — Valley Laser Eye Centre
Locations (1):
- Valley Laser Eye Centre, Abbotsford, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No